CLINICAL TRIAL: NCT01549288
Title: Evaluation of the Modified Atkins Diet in Children With Infantile Spasms Refractory to Hormonal Therapy: a Randomized Controlled Trial
Brief Title: Trial of the Modified Atkins Diet in Infantile Spasms Refractory to Hormonal Therapy
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Satinder Aneja, Assistant Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADIS
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Infantile Spasms
MeSH Terms: conditions — Spasms, Infantile

ARMS (2):
- modified Atkins diet (Experimental)
  Interventions: Behavioral: modified Atkins diet
- control arm (Other): the control arm continues the anti-epileptic drugs without any added dietetic input
  Interventions: Other: no dietetic input

INTERVENTIONS:
Behavioral: modified Atkins diet — Carbohydrate restricted to 10 g/day (18-36 months) and 5 g/day (9-18 months), fat intake encouraged, proteins unrestricted
  Arms: modified Atkins diet
Other: no dietetic input — continuation of anti-epileptic medication without any dietetic input
  Arms: control arm

SUMMARY:
Infantile spasms comprise an infantile epileptic encephalopathy characterized by hypsarrhythmia on EEG, and frequent neurodevelopmental regression. Unfortunately the treatment of this disorder remains difficult. The first-line options which include hormonal therapy, i.e., adrenocorticotropic hormone (ACTH) or oral corticosteroids, and vigabatrin are effective in 60-70% of the patients. Hormonal therapy is considered the best available treatment. Vigabatrin being expensive and of limited availability is not a feasible option for most patients in our setting. Also, these are however associated with significant side effects, and high relapse rates. Newer drugs such as topiramate, zonisamide, and levetiracetam have also been evaluated; however these drugs are less effective than ACTH. The ketogenic diet (KD) is a high fat, low carbohydrate diet. It has been used for treatment of intractable childhood epilepsy. The KD has also been shown to be effective for intractable infantile spasms; often after ACTH and vigabatrin have failed.

The modified Atkins diet is a non-pharmacologic therapy for intractable childhood epilepsy that was designed to be a less restrictive alternative to the traditional ketogenic diet. This diet is started on an outpatient basis without a fast, allows unlimited protein and fat, and does not restrict calories or fluids. Preliminary data have shown efficacy in refractory infantile spasms. This diet is also ideal for resource-constraint settings with paucity of trained dieticians. Hence this study has been planned to evaluate the efficacy and tolerability of the modified Atkins diet in children with infantile spasms refractory to hormonal treatment in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. age 9 months to 3 years
2. Presence of epileptic spasms in clusters in child 9 months to < 3years of age, with electroencephalographic evidence of hypsarrhythmia or its variants), persisting, at least one cluster per day, despite treatment with either oral corticosteroids or adrenocorticotrophic hormone (ACTH) and one additional anticonvulsant (valproate/benzodiazepine/vigabatrin/topiramate/zonisamide/ levetiracetam) for at least 4 weeks.

Exclusion Criteria:

* Children with known or suspected inborn error of metabolism, Patients with clinical suspicion of metabolic disorder as evidenced by 2 or more of the following:

  * a history of parental consanguinity,
  * prior affected siblings,
  * unexplained vomiting,
  * intermittent worsening of symptoms,
  * recurrent episodes of lethargy,
  * altered sensorium, or
  * ataxia,
  * hepatosplenomegaly on examination
* With or without 2 or more of the following biochemical abnormalities:

  * High blood ammonia (> 80mmol/L),
  * High arterial lactate (> 2 mmol/L),
  * metabolic acidosis (pH < 7.2),
  * hypoglycaemia (blood sugar < 40 mg/dl),
  * abnormal urinary aminoacidogram,
  * presence of reducing sugars or ketones in urine, and
  * positive results on urine neurometabolic screening tests. In such patients, blood tandem mass spectrometry or urine gas chromatography mass spectroscopy (GCMS) will be obtained to look for inborn error of metabolism.
* Children with renal, pulmonary, cardiac or hepatic dysfunction
* Severe malnutrition (weight for length and height for age less than 3 SD for mean as per WHO growth charts),
* Children from families who lack motivation will also be excluded as it might affect the compliance.

Ages: 9 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of children who achieved spasm freedom as per parental reports at 4 weeks | 4 weeks

SECONDARY OUTCOMES:
Proportion of children who achieved >50% reduction of clinical spasm, as per parental reports at 4 weeks | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Hardinge Medical College and Associated Kalawati Saran Children's Hospital, New Delhi, National Capital Territory of Delhi, India